CLINICAL TRIAL: NCT01439659
Title: A Randomized Phase II Study of the Nutritional Supplements Juice Plus + and Juice Plus + Complete in Ovarian Cancer Patients
Brief Title: Juice Plus+ and Juice Plus+ Complete in Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Natural Alternatives International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID00-420; NCI-2011-03303 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Epithelial ovarian cancer; First clinical remission; Nutritional Supplements; Juice Plus +; Juice Plus + Complete; Dietary counseling
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional Counseling (Other): For 6 months control group receives dietary counseling.
  Interventions: Behavioral: Nutritional Counseling
- Daily Supplements (Experimental): 2 capsules (Juice Plus+) twice a day (morning and evening) plus Juice Plus+ Complete drink each evening for 6 months.
  Interventions: Dietary Supplement: Daily Supplements

INTERVENTIONS:
Behavioral: Nutritional Counseling — Initial interview and subsequent telephone contact once per week for two months, once every other week for the following two months, and once per month for the remaining two months.
  Arms: Nutritional Counseling
Dietary Supplement: Daily Supplements — Two capsules daily in the morning and two capsules daily in the evening of Juice Plus+ in addition to regular meal. Also a beverage, Juice Plus+ Complete (a powder mixture to be added to one cup of fluid) daily in the evening.
  Arms: Daily Supplements

SUMMARY:
The goal of this clinical research study is to see if ovarian cancer patients who add Juice PLus+ and Juice Plus+ Complete to their diets have better outcomes when compared to ovarian cancer patients who receive only dietary counseling alone.

DETAILED DESCRIPTION:
Before starting the study, patients will have a dietary pattern evaluation, physical exam, blood test, height, weight, hip, wrist, mid-arm and waist circumference measurements.

Researchers will compare changes in weight, waist, hip, mid-arm and wrist size, and changes in the amount of vitamins, iron, and nutrients in the blood. Researchers will also measure the levels of some proteins that can be linked to ovarian tumors.

Patients will be randomly picked (as in the toss of a coin) to be in one of two groups. One group will receive free of charge nutritional counseling for 6 months, while the second group will receive free of charge daily supplements . These supplements will be made up of a combination from fruits and vegetables (Juice Plus+). Patients will be asked to take two capsules (Juice Plus+) in the morning, and two capsules (Juice Plus+) along with a drink containing vitamins and minerals (Juice Plus+ Complete) in the evening for 6 months.

All patients will have their eating patterns monitored for six months. Patients will come to the clinic at least every three months as part of their normal treatment schedule. Each visit will take 3 hours and will include a physical exam, blood tests, and anthropometric measurements (height, weight, waist, hip, mid-arm, and wrist circumferences). At some visits, dietary and quality of life assessments will also be done.

With the exception of the first interview, nutritional counseling will be mostly done by a 30 to 60 minute telephone call once a week for two months. Counseling will also be done once every other week for two months and then once a month for two months.

Participation in this study will be stopped if patients have to start being fed by vein, patients get pregnant or begin breast feeding, patients have bowel obstruction, patients are diagnosed with a condition requiring a restricted diet, patients begin medication that is incompatible with a high fiber diet, or patients have severe side effects.

This is an investigational study. A total of 50 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) > 19.5
2. Epithelial ovarian cancer of (any tumor type). Stages 2 and up.
3. In first clinical remission. (CA125 < 35)
4. > 21 years of age.
5. CT scan of abdomen/pelvis without evidence of ovarian cancer.
6. Ambulatory/mobile and able to eat/not on parenteral nutrition.
7. Life expectancy of at least 6 months.
8. Informed consent signed indicating patient's knowledge of the investigational nature of the study.

Exclusion Criteria:

1. Evidence of bowel obstruction.
2. Pregnant or lactating.
3. Diagnosed with a co-morbidity requiring a restricted diet or medication for which a high fiber diet may be contraindicated.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2003-02-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum lipid peroxide levels resulting from nutritional supplements or dietary counseling | Baseline to 6 months
  Measurements of serum lipid peroxide and serum carotenoid levels obtained at baseline and at least every 3 months for total of 6 months; 3 measurements per participant used to assess changes in the lipid peroxide and serum carotenoid levels - baseline measurement during and after treatment. Outcome evaluated using repeated measures ANOVA design with 2 groups and 3 time points.
Change in levels of serum carotenoid resulting from nutritional supplements or dietary counseling | Baseline to 6 months
  Measurements of serum lipid peroxide and serum carotenoid levels obtained at baseline and at least every 3 months for total of 6 months; 3 measurements per participant used to assess changes in the lipid peroxide and serum carotenoid levels - baseline measurement during and after treatment. Outcome evaluated using repeated measures ANOVA design with 2 groups and 3 time points.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly C. Handy, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org